CLINICAL TRIAL: NCT02927535
Title: Evaluation of TNFα Blockers Monotherapy in Early Rheumatoid Arthritis in France
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Bourse TNFblockers monotherapy
Record Dates: First submitted 2016-09-16; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: TNF blockers monotherapy

SUMMARY:
Aim: To describe 1) The use of TNF blockers monotherapy in early arthritis in daily clinical practice in France 2) To evaluate symptomatic, structural efficacy, and retention rate over 5 years of TNF blockers monotherapy 3) To evaluate predictive factors for TNF blocker response monotherapy Type of study: Observational cohort study using cross-section and longitudinal data.

Description of the project methodology

* Patients: All patients in the ESPOIR cohort (multicentre French cohort study of early RA).A sub-analysis will be conducted among patients satisfying the ACR-EULAR 2010 criteria.
* Data collected: Patient characteristics, Clinical data regarding RA and related pathologies, Characteristics of treatments received The analysis will be conducted using data collected at baseline, 6, 12, 18, 24, 36, 48, 60 months.
* Analyses:

  1. Frequency of use of TNF blockers monotherapy: we will calculate the % of patients initiating TNF blockers monotherapy (Kaplan-Meier method), and we will describe the type of TNF blocker, the route of administration, the dosage, and the place of the TNF blockers monotherapy in the treatment strategy during the first 5 years.
  2. Identification of potential predictive factors for initiation of TNF blockers monotherapy: a survival curve (Kaplan-Meier) will be performed. The baseline characteristics of the patients with regard to the initiation of TNF blocker monotherapy during the first 5 years of the disease will be compared by univariate analysis and Log-rank test will be performed in all variables. A stepwise multivariate analysis (Cox analysis) will be performed.
  3. Therapeutical effect: we will calculate the retention rate over time, and will compare the changes in different variables in the group of patients who have received TNF blockers monotherapy matched (using a propensity score) to 1,2 or 3 patients who have received TNF blockers in combination with synthetic DMARDs. We will assess and compare DAS28 and HAQ at short term (after at least 8 weeks of treatment) and long term (last available visit) in groups. The structural efficacy was evaluated by the radiographic progression at last available visit. We will identically estimate the drug effect depending on the TNF blocker used, by calculating the retention rate and comparing DAS28 at short term and long term.
  4. Identification of predictive factors for TNF blocker monotherapy response: To evaluate the impact of baseline demographics and disease conditions on the DAS28 and HAQ response during the first 5 years will be compared by univariate and multivariate analysis.

Expected results:

Increase knowledge on the use of TNF blocker monotherapy, its efficacy and retention rate, and on predictive factors for TNF blocker monotherapy response in early RA patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 70 years
* more than 2 swollen joints for >6 weeks and <6 months
* suspected or confirmed diagnosis of RA
* no previous intake of DMARDs or steroids (except if <2 weeks).

Exclusion Criteria:

* Patients were excluded if the referring physician judged they had other clearly defined inflammatory rheumatic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the ESPOIR cohort (multicentre French cohort study of early RA). A sub-analysis will be conducted among patients satisfying the ACR-EULAR 2010 criteria.
Sampling Method: Non-Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Frequency of use of TNF blocker monotherapy | baseline (day 0)
Frequency of use of TNF blocker monotherapy | 6 months
Frequency of use of TNF blocker monotherapy | 12 months
Frequency of use of TNF blocker monotherapy | 18 months
Frequency of use of TNF blocker monotherapy | 24 months
Frequency of use of TNF blocker monotherapy | 36 months
Frequency of use of TNF blocker monotherapy | 48 months
Frequency of use of TNF blocker monotherapy | 60 months
Frequency of use of TNF blocker monotherapy | 120 months